CLINICAL TRIAL: NCT01449812
Title: Immunogenicity and Safety of a Booster Dose of GlaxoSmithKline Biologicals' IPV (Poliorix™) and DTPa/Hib (Infanrix+Hib™) in Healthy Chinese Toddlers
Brief Title: Immunogenicity and Safety Study of Booster Dose of GSK Biologicals' IPV (Poliorix™) and DTPa/Hib (Infanrix+Hib™) Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 114386
Record Dates: First submitted 2011-10-06; First posted 2011-10-10 (Estimated); Results first posted 2017-04-13 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2017-04

CONDITIONS: Acellular Pertussis; Tetanus; Diphtheria; Haemophilus Influenzae Type b
Keywords: combination vaccine; booster vaccination
MeSH Terms: conditions — Tetanus; Diphtheria; Haemophilus Infections | interventions — diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine; Pentetic Acid

ARMS (3):
- INFANRIX+HIB/POLIORIX 1 GROUP (Experimental): Healthy male or female children between, and including, 18 and 24 months of age at the time of booster vaccination, who were primed with 3 doses of the Infanrix-IPV/Hib™ vaccine at 2, 3 and 4 months of age in the DTPA-IPV-056 (112584) primary study, additionally received 1 dose of Poliorix™ and of Infanrix+Hib™ vaccines, administered intramuscularly into the upper sides of the left and right thighs, respectively.
  Interventions: Biological: Infanrix+Hib™; Biological: Poliorix™
- INFANRIX+HIB/POLIORIX 2 GROUP (Experimental): Healthy male or female children between, and including, 18 and 24 months of age at the time of booster vaccination, who were primed with 3 doses of the Infanrix-IPV/Hib™ vaccine at 3, 4 and 5 months of age in the DTPA-IPV-056 (112584) primary study, additionally received 1 dose of Poliorix™ and of Infanrix+Hib™ vaccines, administered intramuscularly into the upper sides of the left and right thighs, respectively.
  Interventions: Biological: Infanrix+Hib™; Biological: Poliorix™
- CONTROL GROUP (Active Comparator): Healthy male or female children between, and including, 18 and 24 months of age at the time of booster vaccination, who were primed with 3 doses of the Infanrix+Hib™ and of Poliorix™ vaccines at 2, 3 and 4 months of age in the DTPA-IPV-056 (112584) primary study, additionally received 1 dose of Poliorix™ and of Infanrix+Hib™ vaccines, administered intramuscularly into the upper sides of the left and right thighs, respectively.
  Interventions: Biological: Infanrix+Hib™; Biological: Poliorix™

INTERVENTIONS:
Biological: Infanrix+Hib™ — Intramuscular, one dose
  Other Names: DTPa /Hib
Biological: Poliorix™ — Intramuscular, one dose
  Other Names: IPV

SUMMARY:
The purpose of this booster study is to evaluate the immune persistence in healthy Chinese subjects primed in study NCT01086423 with GSK Biologicals' Infanrix-IPV+Hib™ (DTPa-IPV/Hib) vaccine. The study will also evaluate the safety and immune response of these subjects to a booster dose of Infanrix-Hib™ (DTPa/Hib) and Poliorix™ (IPV) vaccine.

This protocol posting deals with objectives & outcome measures of the booster phase. The objectives & outcome measures of the primary phase are presented in a separate protocol posting (NCT number = NCT01086423).

ELIGIBILITY:
Inclusion Criteria:

* A male or female child between, and including, 18 and 24 months of age at the time of the booster vaccination.
* Subjects who completed the full three-dose primary vaccination course in study NCT01086423.
* Subjects who the investigator believes that their parent(s)/ Legally Acceptable Representative(s) LAR(s) can and will comply with the requirements of the protocol
* Written informed consent obtained from the parent(s)/LAR(s) of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Child in care
* Use of any investigational or non-registered product other than the study vaccine(s) within 30 days preceding the booster dose of the study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the booster dose.
* Administration of a vaccine not foreseen by the study protocol within 30 days prior to the booster vaccination, or planned administration during the study period.
* Participation in another clinical study within three months prior to enrolment in the present booster study or at any time during the present booster study, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Evidence of previous diphtheria, tetanus, pertussis, poliomyelitis and Haemophilus influenzae type b, vaccination or disease since the conclusion visit of primary study NCT01086423.
* Serious chronic illness.
* Administration of immunoglobulins and/or any blood products within the 90 days preceding the booster dose of study vaccine or planned administration during the study period.
* Occurrence of any of the following adverse events after a previous administration of a DTP vaccine.
* Encephalopathy
* Temperature of ≥ 40.0°C (axillary temperature) within 48 hours of vaccination, not due to another identifiable cause.
* Collapse or shock-like state within 48 hours of vaccination.
* Persistent, inconsolable crying occurring within 48 hours of vaccination and lasting ≥ 3 hours.
* Seizures with or without fever occurring within 3 days of vaccination.

The following condition is temporary or self-limiting, and a subject may be vaccinated once the condition has resolved if no other exclusion criteria is met:

* Acute disease and/or fever at the time of enrolment.

Ages: 18 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 831 (Actual)
Dates: Start 2011-10-01; Primary Completion 2012-01-16 (Actual); Study Completion 2012-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Wuzhou, Guangxi, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 6 subjects did not receive vaccination.
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Period: Overall Study
Arm/Group | Infanrix+Hib/Poliorix 1 Group | Infanrix+Hib/Poliorix 2 Group | Control Group
Started | 272 | 273 | 280
Completed | 270 | 273 | 279
Not Completed | 2 | 0 | 1
Not completed — Migrated/moved from study area | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Infanrix+Hib/Poliorix 1 Group | Infanrix+Hib/Poliorix 2 Group | Control Group | Total
Number analyzed (Participants) | 272 | 273 | 280 | 825
Age, Continuous [Mean (Standard Deviation); unit: Months] | 19.5 (0.93) | 19.4 (0.91) | 19.5 (0.97) | 19.47 (0.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 131 | 126 | 120 | 377
  Male | 141 | 147 | 160 | 448
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian-Chinese heritage | 272 | 273 | 280 | 825

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroprotected Subjects Against Diphtheria (D) and Tetanus (T) Toxoids
Description: A seroprotected subject was defined as a vaccinated subject with anti-D and anti-T antibody concentrations greater than or equal to (≥) 0.1 international units per milliliter (IU/mL).
Time Frame: Before the booster vaccination (At Day 0)
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for analysis of antibody persistence, which included all subjects who have completed their full three-dose primary vaccination course in the DTPA-IPV-056 study and for whom serological results were available at the persistence time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix+Hib/Poliorix 1 Group | Infanrix+Hib/Poliorix 2 Group | Control Group
Number analyzed (Participants) | 272 | 273 | 279
Participants
  Anti-D: number analyzed (Participants) | 271 | 272 | 279
  Anti-D | 241 | 250 | 234
  Anti-T: number analyzed (Participants) | 272 | 273 | 278
  Anti-T | 269 | 271 | 275

2. Primary Outcome: Anti-D and Anti-T Antibody Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs) for the seroprotection cut-off of ≥0.1 IU/mL.
Time Frame: Before the booster vaccination (At Day 0)
Population: The analysis was performed on the ATP cohort for analysis of antibody persistence, which included all subjects who have completed their full three-dose primary vaccination course in the DTPA-IPV-056 study and for whom serological results were available at the persistence time point.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Infanrix+Hib/Poliorix 1 Group | Infanrix+Hib/Poliorix 2 Group | Control Group
Number analyzed (Participants) | 272 | 273 | 279
IU/mL
  Anti-D: number analyzed (Participants) | 271 | 272 | 279
  Anti-D | 0.175 [0.163 to 0.188] | 0.189 [0.176 to 0.202] | 0.154 [0.142 to 0.166]
  Anti-T: number analyzed (Participants) | 272 | 273 | 278
  Anti-T | 0.45 [0.423 to 0.478] | 0.509 [0.481 to 0.54] | 0.38 [0.359 to 0.404]

3. Primary Outcome: Number of Seroprotected Subjects Against Polyribosyl-ribitol-phosphate (Anti-PRP)
Description: A seroprotected subject was defined as a vaccinated subject with anti-PRP antibody concentration ≥ 0.15 micrograms per milliliter (µg/mL).
Time Frame: Before the booster vaccination (At Day 0)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix+Hib/Poliorix 1 Group | Infanrix+Hib/Poliorix 2 Group | Control Group
Number analyzed (Participants) | 272 | 273 | 280
Participants | 226 | 234 | 241

4. Primary Outcome: Anti-PRP Antibody Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs) for the seroprotection cut-off of ≥ 0.15 µg/mL.
Time Frame: Before the booster vaccination (At Day 0)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Infanrix+Hib/Poliorix 1 Group | Infanrix+Hib/Poliorix 2 Group | Control Group
Number analyzed (Participants) | 272 | 273 | 280
µg/mL | 2.275 [1.856 to 2.788] | 2.674 [2.193 to 3.26] | 2.413 [2.006 to 2.904]

5. Primary Outcome: Number of Seroprotected Subjects Against Polio Type 1, 2 and 3
Description: A seroprotected subject was defined as a vaccinated subject with anti-polio type 1, 2 and 3 antibody concentrations ≥ the cut-off value of 8 Estimated Dose 50% (ED50). ED50 is the estimated serum dilution reducing the signal generated by viral infection with 50%.
Time Frame: Before the booster vaccination (At Day 0)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix+Hib/Poliorix 1 Group | Infanrix+Hib/Poliorix 2 Group | Control Group
Number analyzed (Participants) | 272 | 273 | 280
Participants
  Anti-polio 1 | 259 | 267 | 270
  Anti-polio 2 | 248 | 261 | 250
  Anti-polio 3 | 254 | 259 | 257

6. Primary Outcome: Anti-polio Type 1, 2 and 3 Antibody Titers
Description: Antibody titers were presented as geometric mean titers (GMTs) for the seroprotection cut-off of ≥ 8.
Time Frame: Before the booster vaccination (At Day 0)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Infanrix+Hib/Poliorix 1 Group | Infanrix+Hib/Poliorix 2 Group | Control Group
Number analyzed (Participants) | 272 | 273 | 280
Titers
  Anti-polio 1 | 72.3 [62.4 to 83.7] | 95.7 [82.5 to 111] | 77.2 [67 to 89]
  Anti-polio 2 | 57.3 [47 to 70] | 63.6 [53.5 to 75.5] | 42.6 [35.7 to 50.8]
  Anti-polio 3 | 71.3 [60.1 to 84.7] | 79.9 [66.4 to 96.2] | 60.6 [51.2 to 71.8]

7. Primary Outcome: Number of Seropositive Subjects for Anti-pertussis Toxoid (Anti-PT), Anti-filamentous Haemagglutinin (Anti-FHA) and Anti-pertactin (Anti-PRN)
Description: A seropositive subject was defined as a vaccinated subject with anti-PT, anti-FHA and anti-PRN antibody concentration ≥ 5 enzyme-linked immunosorbent assay (ELISA) units per milliliter (EL.U/ml).
Time Frame: Before the booster vaccination (At Day 0)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix+Hib/Poliorix 1 Group | Infanrix+Hib/Poliorix 2 Group | Control Group
Number analyzed (Participants) | 272 | 273 | 280
Participants
  Anti-PT | 260 | 263 | 260
  Anti-FHA | 262 | 267 | 262
  Anti-PRN | 260 | 265 | 267

8. Primary Outcome: Anti-PT, Anti-FHA and Anti-PRN Antibody Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs) for the seropositivity cut-off of ≥ 5 EL.U/mL.
Time Frame: Before the booster vaccination (At Day 0)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Infanrix+Hib/Poliorix 1 Group | Infanrix+Hib/Poliorix 2 Group | Control Group
Number analyzed (Participants) | 272 | 273 | 280
EL.U/mL
  Anti-PT | 10.3 [9.6 to 11.1] | 12.2 [11.3 to 13.1] | 10.4 [9.6 to 11.2]
  Anti-FHA | 12.8 [11.9 to 13.7] | 14.3 [13.4 to 15.2] | 12.4 [11.5 to 13.4]
  Anti-PRN | 9.2 [8.8 to 9.7] | 9.7 [9.2 to 10.1] | 9 [8.5 to 9.5]

9. Primary Outcome: Number of Seroprotected Subjects Against Diphteria (D) and Tetanus (T) Toxoids
Description: A seroprotected subject was defined as a vaccinated subject with anti-D and anti-T antibody concentrations greater than or equal to (≥) 0.1 IU/mL.
Time Frame: Before the booster vaccination (At Day 0)
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome measures and assay results for antibodies against at least one study vaccine antigen component after vaccination were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix+Hib/Poliorix 1 Group | Infanrix+Hib/Poliorix 2 Group | Control Group
Number analyzed (Participants) | 266 | 268 | 272
Participants
  Anti-D: number analyzed (Participants) | 265 | 267 | 272
  Anti-D | 235 | 245 | 228
  Anti-T: number analyzed (Participants) | 266 | 268 | 271
  Anti-T | 264 | 266 | 268

10. Primary Outcome: Number of Seroprotected Subjects Against Diphteria (D) and Tetanus (T) Toxoids
Description: A seroprotected subject was defined as a vaccinated subject with anti-D and anti-T antibody concentrations ≥ 0.1 IU/mL.
Time Frame: One month after the booster vaccination (At Month 1)
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome measures and assay results for antibodies against at least one study vaccine antigen component after vaccination were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix+Hib/Poliorix 1 Group | Infanrix+Hib/Poliorix 2 Group | Control Group
Number analyzed (Participants) | 266 | 268 | 272
Participants
  Anti-D: number analyzed (Participants) | 265 | 268 | 270
  Anti-D | 265 | 268 | 270
  Anti-T | 266 | 268 | 272

11. Primary Outcome: Anti-D and Anti-T Antibody Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs) for the seroprotection cut-off of ≥ 0.1 IU/mL.
Time Frame: Before the booster vaccination (At Day 0)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Infanrix+Hib/Poliorix 1 Group | Infanrix+Hib/Poliorix 2 Group | Control Group
Number analyzed (Participants) | 266 | 268 | 272
IU/mL
  Anti-D: number analyzed (Participants) | 265 | 267 | 272
  Anti-D | 0.174 [0.162 to 0.187] | 0.189 [0.176 to 0.202] | 0.154 [0.142 to 0.166]
  Anti-T: number analyzed (Participants) | 266 | 268 | 271
  Anti-T | 0.455 [0.429 to 0.483] | 0.511 [0.482 to 0.542] | 0.38 [0.357 to 0.403]

12. Primary Outcome: Anti-D and Anti-T Antibody Concentrations
Description: Antibody concentrations were presented as GMCs for the seroprotection cut-off of ≥ 0.1 IU/mL.
Time Frame: One month after the booster vaccination (At Month 1)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Infanrix+Hib/Poliorix 1 Group | Infanrix+Hib/Poliorix 2 Group | Control Group
Number analyzed (Participants) | 266 | 268 | 272
IU/mL
  Anti-D: number analyzed (Participants) | 265 | 268 | 270
  Anti-D | 1.341 [1.239 to 1.451] | 1.504 [1.377 to 1.643] | 1.227 [1.134 to 1.326]
  Anti-T | 4.862 [4.614 to 5.124] | 4.927 [4.693 to 5.173] | 4.371 [4.161 to 4.591]

13. Primary Outcome: Number of Seroprotected Subjects Against Polyribosyl-ribitol-phosphate (PRP)
Description: A seroprotected subject was defined as a vaccinated subject with anti-PRP antibody concentration ≥ 0.15 µg/mL.
Time Frame: Before the booster vaccination (At Day 0)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix+Hib/Poliorix 1 Group | Infanrix+Hib/Poliorix 2 Group | Control Group
Number analyzed (Participants) | 266 | 268 | 273
Participants | 221 | 229 | 234

14. Primary Outcome: Number of Seroprotected Subjects Against PRP
Description: A seroprotected subject was defined as a vaccinated subject with anti-PRP antibody concentrations ≥ 0.15 µg/mL.
Time Frame: One month after the booster vaccination (At Month 1)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix+Hib/Poliorix 1 Group | Infanrix+Hib/Poliorix 2 Group | Control Group
Number analyzed (Participants) | 266 | 268 | 273
Participants | 264 | 268 | 271

15. Primary Outcome: Anti-PRP Antibody Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs) for the seroprotection cut-off of ≥ 0.15 micrograms per milliliter (µg/mL).
Time Frame: Before the booster vaccination (At Day 0)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Infanrix+Hib/Poliorix 1 Group | Infanrix+Hib/Poliorix 2 Group | Control Group
Number analyzed (Participants) | 266 | 268 | 273
µg/mL | 2.308 [1.878 to 2.836] | 2.743 [2.245 to 3.352] | 2.407 [1.993 to 2.908]

16. Primary Outcome: Anti-PRP Antibody Concentrations
Description: as for outcome 4
Time Frame: One month after the booster vaccination (At Month 1)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Infanrix+Hib/Poliorix 1 Group | Infanrix+Hib/Poliorix 2 Group | Control Group
Number analyzed (Participants) | 266 | 268 | 273
µg/mL | 35.178 [30.617 to 40.418] | 49.023 [43.649 to 55.058] | 27.682 [24.251 to 31.598]

17. Primary Outcome: Number of Seroprotected Subjects for Anti-polio Type 1, 2 and 3
Description: A seroprotected subject was defined as a vaccinated subject with anti-polivirus antibody concentration ≥ 8 ED50. ED50 is the estimated serum dilution reducing the signal generated by viral infection with 50%.
Time Frame: Before the booster vaccination (At Day 0)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix+Hib/Poliorix 1 Group | Infanrix+Hib/Poliorix 2 Group | Control Group
Number analyzed (Participants) | 266 | 268 | 273
Participants
  Anti-Polio 1 | 253 | 262 | 263
  Anti-Polio 2 | 243 | 256 | 244
  Anti-Polio 3 | 249 | 254 | 250

18. Primary Outcome: Number of Seroprotected Subjects Against Polio Type 1, 2 and 3
Description: A seroprotected subject was defined as a vaccinated subject with anti-polivirus antibody concentrations ≥ 8 ED50. ED50 is the estimated serum dilution reducing the signal generated by viral infection with 50%.
Time Frame: One month after the booster vaccination (At Month 1)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix+Hib/Poliorix 1 Group | Infanrix+Hib/Poliorix 2 Group | Control Group
Number analyzed (Participants) | 265 | 268 | 273
Participants
  Anti-Polio 1 | 265 | 268 | 273
  Anti-Polio 2 | 265 | 268 | 273
  Anti-Polio 3 | 265 | 268 | 273

19. Primary Outcome: Anti-polio Type 1, 2 and 3 Antibody Titers
Description: Antibody titers were presented as geometric mean titers (GMTs) for the seroprotection cut-off of ≥ the value of 8.
Time Frame: Before the booster vaccination (At Day 0)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Infanrix+Hib/Poliorix 1 Group | Infanrix+Hib/Poliorix 2 Group | Control Group
Number analyzed (Participants) | 266 | 268 | 273
Titers
  Anti-Polio 1 | 72 [62 to 83.7] | 96.3 [82.8 to 112] | 75.9 [65.7 to 87.6]
  Anti-Polio 2 | 56.5 [46.2 to 69] | 64.1 [53.8 to 76.4] | 41.9 [35 to 50]
  Anti-Polio 3 | 72.6 [61.1 to 86.3] | 79.4 [65.8 to 95.8] | 60.3 [50.8 to 71.6]

20. Primary Outcome: Anti-polio Type 1, 2 and 3 Antibody Titers
Description: Antibody titers were presented as geometric mean titers (GMTs) for the seroprotection cut-off of ≥ 8.
Time Frame: One month after the booster vaccination (At Month 1)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Infanrix+Hib/Poliorix 1 Group | Infanrix+Hib/Poliorix 2 Group | Control Group
Number analyzed (Participants) | 265 | 268 | 273
Titers
  Anti-Polio 1 | 3512.2 [3159.7 to 3904.1] | 3410.9 [3081.7 to 3775.4] | 3386.8 [3078 to 3726.6]
  Anti-Polio 2 | 1931.2 [1721.7 to 2166.2] | 2237.9 [2001.6 to 2502.1] | 1886.1 [1679.6 to 2117.9]
  Anti-Polio 3 | 5237.8 [4671.8 to 5872.3] | 5438.5 [4846.8 to 6102.4] | 5141.2 [4650.1 to 5684.2]

21. Primary Outcome: Number of Seropositive Subjects for Anti-PT, Anti-FHA and Anti-PRN
Description: A seropositive subject was defined as a vaccinated subject with anti-PT, anti-FHA and anti-PRN antibody concentrations ≥ 5 ELISA units per milliliter (EL.U/mL).
Time Frame: Before the booster vaccination (At Day 0)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix+Hib/Poliorix 1 Group | Infanrix+Hib/Poliorix 2 Group | Control Group
Number analyzed (Participants) | 266 | 268 | 273
Participants
  Anti-PT | 254 | 258 | 253
  Anti-FHA | 256 | 262 | 255
  Anti-PRN | 254 | 260 | 260

22. Primary Outcome: Number of Seropositive Subjects for Anti-PT, Anti-FHA and Anti-PRN
Description: A seropositive subject was defined as a vaccinated subject with anti-PT, anti-FHA and anti-PRN antibody concentrations ≥ 5 EL.U/mL.
Time Frame: One month after the booster vaccination (At Month 1)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix+Hib/Poliorix 1 Group | Infanrix+Hib/Poliorix 2 Group | Control Group
Number analyzed (Participants) | 266 | 268 | 273
Participants
  Anti-PT | 266 | 268 | 273
  Anti-FHA | 266 | 268 | 273
  Anti-PRN | 266 | 268 | 273

23. Primary Outcome: Anti-PT, Anti-FHA and Anti-PRN Antibody Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs) for the seropositivity cut-off value of ≥ 5 EL.U/mL.
Time Frame: Before the booster vaccination (At Day 0)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Infanrix+Hib/Poliorix 1 Group | Infanrix+Hib/Poliorix 2 Group | Control Group
Number analyzed (Participants) | 266 | 268 | 273
EL.U/mL
  Anti-PT | 10.3 [9.5 to 11.1] | 12.2 [11.3 to 13.1] | 10.3 [9.5 to 11.2]
  Anti-FHA | 12.7 [11.8 to 13.6] | 14.3 [13.4 to 15.2] | 12.3 [11.4 to 13.3]
  Anti-PRN | 9.2 [8.7 to 9.6] | 9.7 [9.2 to 10.2] | 9 [8.5 to 9.5]

24. Primary Outcome: Anti-PT, Anti-FHA and Anti-PRN Antibody Concentrattions
Description: as for outcome 8
Time Frame: One month after the booster vaccination (At Month 1)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Infanrix+Hib/Poliorix 1 Group | Infanrix+Hib/Poliorix 2 Group | Control Group
Number analyzed (Participants) | 266 | 268 | 273
EL.U/mL
  Anti-PT | 138.5 [132 to 145.3] | 146.2 [139.7 to 153] | 126.8 [120.4 to 133.5]
  Anti-FHA | 124.6 [119.2 to 130.2] | 124 [119.2 to 129] | 120.8 [115.3 to 126.6]
  Anti-PRN | 57.3 [55.6 to 59.1] | 59.9 [58.1 to 61.8] | 57.2 [55.3 to 59.1]

25. Primary Outcome: Number of Subjects With a Booster Response to Anti-PT, Anti-FHA and Anti-PRN
Description: Booster response was defined as the appearance of antibodies in subjects who were initially seronegative (i.e. with concentrations < cut-off value) or at least maintenance of pre-vaccination antibody concentrations in subjects who were initially seropositive (i.e. with concentrations ≥ cut-off value), taking into consideration the decreasing maternal antibodies.
Time Frame: One month after the booster vaccination (At Month 1)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix+Hib/Poliorix 1 Group | Infanrix+Hib/Poliorix 2 Group | Control Group
Number analyzed (Participants) | 266 | 268 | 273
Participants
  Anti-PT | 266 | 268 | 272
  Anti-FHA | 266 | 268 | 272
  Anti-PRN | 239 | 230 | 244

26. Secondary Outcome: Number of Subjects With Any Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade.
Time Frame: During the 4-day (Days 0-3) post-vaccination period
Population: The analysis was performed on the Total Vaccinated Cohort, which included all subjects with the symptoms sheet filled in, who had received the booster dose and for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix+Hib/Poliorix 1 Group | Infanrix+Hib/Poliorix 2 Group | Control Group
Number analyzed (Participants) | 270 | 273 | 279
Participants
  Any Pain | 73 | 74 | 76
  Any Redness | 19 | 15 | 19
  Any Swelling | 16 | 10 | 14

27. Secondary Outcome: Number of Subjects With Any Solicited General Symptoms
Description: Assessed solicited general symptoms were drowsiness, irritability, loss of appetite and fever [defined as axillary temperature equal to or above 37.1 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade and relationship to vaccination.
Time Frame: During the 4-day (Days 0-3) post-vaccination period
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix+Hib/Poliorix 1 Group | Infanrix+Hib/Poliorix 2 Group | Control Group
Number analyzed (Participants) | 270 | 273 | 279
Participants
  Any Drowsiness | 38 | 50 | 38
  Any Irritability | 78 | 81 | 72
  Any Loss of appetite | 67 | 73 | 69
  Any Fever | 102 | 105 | 91

28. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 31-day (Days 0-30) post-vaccination period
Population: The analysis was performed on the Total Vaccinated Cohort, which included all subjects who had received the booster dose and for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix+Hib/Poliorix 1 Group | Infanrix+Hib/Poliorix 2 Group | Control Group
Number analyzed (Participants) | 272 | 273 | 280
Participants | 16 | 13 | 21

29. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period (from Month 0 up to Month 1)
Population: as for outcome 28
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix+Hib/Poliorix 1 Group | Infanrix+Hib/Poliorix 2 Group | Control Group
Number analyzed (Participants) | 272 | 273 | 280
Participants | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 4-day (Days 0-3) post-vaccination period. AEs: within the 31-day (Days 0-30) period following booster vaccination. SAEs: throughout the entire study period (from Month 0 up to Month 1).
Arm/Group | Infanrix+Hib/Poliorix 1 Group | Infanrix+Hib/Poliorix 2 Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/272 | 0/273 | 0/280
Serious Adverse Events (participants affected / at risk) | 1/272 | 0/273 | 0/280
Other Adverse Events (participants affected / at risk) | 157/272 | 164/273 | 158/280
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Infanrix+Hib/Poliorix 1 Group (N=272) | Infanrix+Hib/Poliorix 2 Group (N=273) | Control Group (N=280)
Febrile convulsion (Nervous system disorders) | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Infanrix+Hib/Poliorix 1 Group (N=272) | Infanrix+Hib/Poliorix 2 Group (N=273) | Control Group (N=280)
Pain (General disorders) | 73/270 | 74 | 76/279 — This solicited local symptom was only collected from subjects with their symptom sheets completed.
Redness (General disorders) | 19/270 | 15 | 16/279 — This solicited local symptom was only collected from subjects with their symptom sheets completed.
Swelling (General disorders) | 16/270 | 10 | 14/279 — This solicited local symptom was only collected from subjects with their symptom sheets completed.
Drowsiness (General disorders) | 38/270 | 50 | 38/279 — This solicited general symptom was only collected from subjects with their symptom sheets completed.
Irritability (General disorders) | 78/270 | 81 | 72/279 — This solicited general symptom was only collected from subjects with their symptom sheets completed.
Loss of appetite (General disorders) | 67/270 | 73 | 69/279 — This solicited general symptom was only collected from subjects with their symptom sheets completed.
Fever (General disorders) | 102/270 | 105 | 91/279 — This solicited general symptom was only collected from subjects with their symptom sheets completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.